CLINICAL TRIAL: NCT06941701
Title: To Determine the Effects of Physical Fatigue on Cognitive Load and Performance Under Dual-Task Environments.
Brief Title: Effects of Physical Fatigue on Cognitive Load and Performance Under Dual-Task Environments.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: REC/02028 Imran Amjad
Record Dates: First submitted 2025-04-07; First posted 2025-04-24 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Fatigue; Cognitive Load
Keywords: Dual-Task Performance
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Intervention Model Description: Reserach
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Participants with a target Heart rate range of 50-60% of their maximum heart rate. All members of Group 1 who meet the eligibility criteria will perform a cognitive task before undergoing mild-intensity physical fatigue induced by treadmill training. After that participants will complete the cognitive task again. To eliminate bias, three different levels of physical exertion will be randomly assigned.
  Interventions: Other: Mild-intensity physical fatigue
- Group 2 (Experimental): Participants with a target Heart rate range of 60-70% of their maximum heart rate. All members of group 2 who meet the eligibility criteria will perform a cognitive task before undergoing moderate-intensity physical fatigue induced by treadmill training. After that participants will complete the cognitive task again. To eliminate bias, three different levels of physical exertion will be randomly assigned.
  Interventions: Other: Moderate-intensity physical fatigue
- Group 3 (Experimental): Participants with a target Heart rate range of 70-80% of their maximum heart rate. All members of group 3 who meet the eligibility criteria will perform a cognitive task before undergoing high-intensity physical fatigue induced by treadmill training. After that participants will complete the cognitive task again. To eliminate bias, three different levels of physical exertion will be randomly assigned.
  Interventions: Other: High-intensity physical fatigue

INTERVENTIONS:
Other: Mild-intensity physical fatigue — Participants will undergo mild-intensity physical fatigue through a structured treadmill training protocol. The training will be conducted within a target heart rate range of 50-60% of their maximum heart rate (HRmax), ensuring controlled and consistent exercise intensity. This approach aims to induce mild physiological stress while maintaining safety and feasibility for all participants.
  Arms: Group 1
Other: Moderate-intensity physical fatigue — Participants will undergo Moderate-intensity physical fatigue through a structured treadmill training protocol. The training will be conducted within a target heart rate range of 60-70% of their maximum heart rate (HRmax), ensuring controlled and consistent exercise intensity. This approach aims to induce mild physiological stress while maintaining safety and feasibility for all participants.
  Arms: Group 2
Other: High-intensity physical fatigue — Participants will undergo High-intensity physical fatigue through a structured treadmill training protocol. The training will be conducted within a target heart rate range of 70-80% of their maximum heart rate (HRmax), ensuring controlled and consistent exercise intensity. This approach aims to induce sufficient physiological stress while maintaining safety and feasibility for all participants.
  Arms: Group 3

SUMMARY:
This study aims to determine how different levels of physical fatigue influence cognitive load and performance during dual-task activities.

1. To assess the changes in cognitive task performance under varying levels of physical fatigue.
2. There is an association between cognitive loading and physical fatigue.

DETAILED DESCRIPTION:
Working efficiency in our daily routine is hindered by constant change, urgency, and the demands of sustained efforts, all of which contribute to health and safety problems, and are extremely imprudent of human resources in the workplace, due to which individuals would raise anxiety, causing more attention required for task completion and thereby increasing cognitive load. Cognitive loading refers to the mental effort needed to process information and perform tasks. Physical performance is not only related to physical factors, psychological factors also have the potential to determine physical performance. Mental workload is defined as the difference between the cognitive demand of a particular task and the operator's attention resources. When cognitive demands exceed available resources, mental fatigue can occur, often reflected in decreased motor function and impaired physical performance. Fatigue is recognized as a dimensional phenomenon encompassing cognitive and motor fatigue. It is debatable whether cognitive fatigue is a spontaneous phenomenon or provoked by exertion or whether cognitive fatigue is provoked by cognitive effort or also through physical exercise. Physical fatigue develops more quickly when the brain has to devote resources to highly cognitive tasks. Influence of cognitive load on the dynamics of neurophysiological adjustments during exercise which causes fatigue explained by the interaction of various psychological and neurophysiological factors including higher perceived exertion, greater perturbations of autonomic nervous system activity, and cerebral impairments leading to earlier onset of central fatigue. The brain is like other biological tissue tired out when overused. Since the impact of physical exercise on cognitive functioning is dependent on the characteristics of the physical exercise load. Previous research has demonstrated a small-to-medium negative effect of cognitive exertion on subsequent physical performance. Our study aims to explore the interplay between varying levels of physical fatigue and cognitive performance. Specifically, we will examine how different intensities of physical load affect mental load and associated physiological functions. By investigating these relationships, we seek to provide insights into optimizing performance in dual-task environments, ultimately contributing to better health and efficiency in the workplace.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 to 30 years.
* Physically healthy individuals.
* Willingness to participate in the study.

Exclusion Criteria:

* Cognitive Impairment.
* Neurological injury.
* Cardiac, pulmonary, or inflammatory diseases.
* Mental health conditions include depression and post-traumatic stress disorder.
* Individuals unwilling to participate.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — All male and female healthy students are eligible to participate.
Enrollment: 90 (Estimated)
Dates: Start 2025-04-23 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Heart rate variability | Baseline
  An electrocardiogram (ECG) will be utilized to assess heart rate variability, which will measure the fluctuations in time between heartbeats. Low heart rate variability will indicate increased cognitive load.
Heart rate variability (2nd reading) | Periprocedural
  An electrocardiogram (ECG) will be utilized to assess heart rate variability, which will measure the fluctuations in time between heartbeats. Low heart rate variability will indicate increased cognitive load. 2nd reading will be measured during the cognitive task (without physical fatigue).
Heart rate variability (3rd reading) | Periprocedural
  An electrocardiogram (ECG) will be utilized to assess heart rate variability, which will measure the fluctuations in time between heartbeats. Low heart rate variability will indicate increased cognitive load. 3rd reading will be measured after the cognitive task (without physical fatigue).
Heart rate variability (4rth reading) | Periprocedural
  An electrocardiogram (ECG) will be utilized to assess heart rate variability, which will measure the fluctuations in time between heartbeats. Low heart rate variability will indicate increased cognitive load. 4rth reading will be measured after physical fatigue.
Heart rate variability (5th reading) | Periprocedural
  An electrocardiogram (ECG) will be utilized to assess heart rate variability, which will measure the fluctuations in time between heartbeats. Low heart rate variability will indicate increased cognitive load. The 5th reading will be measured during the cognitive task after physical fatigue.
Heart rate variability (6th reading) | Periprocedural
  An electrocardiogram (ECG) will be utilized to assess heart rate variability, which will measure the fluctuations in time between heartbeats. Low heart rate variability will indicate increased cognitive load. The 6th reading will be measured after the cognitive task, after physical fatigue.
Galvanic skin response | Baseline
  The electrical conductance of the skin, measured by Galvanic Skin Response (GSR), will be influenced by moisture levels resulting from sweat gland activity. A high GSR will typically indicate an increased cognitive load.
Galvanic skin response (2nd reading) | Periprocedural
  The electrical conductance of the skin, measured by Galvanic Skin Response (GSR), will be influenced by moisture levels resulting from sweat gland activity. A high GSR will typically indicate an increased cognitive load. 2nd reading will be measured during the cognitive task (without physical fatigue).
Galvanic skin response (3rd reading) | Periprocedural
  The electrical conductance of the skin, measured by Galvanic Skin Response (GSR), will be influenced by moisture levels resulting from sweat gland activity. A high GSR will typically indicate an increased cognitive load. 3rd reading will be measured after the cognitive task (without physical fatigue).
Galvanic skin response (4rth reading) | Periprocedural
  The electrical conductance of the skin, measured by Galvanic Skin Response (GSR), will be influenced by moisture levels resulting from sweat gland activity. A high GSR will typically indicate an increased cognitive load.4rth reading will be measured after physical fatigue.
Galvanic skin response (5th reading) | Periprocedural
  The electrical conductance of the skin, measured by Galvanic Skin Response (GSR), will be influenced by moisture levels resulting from sweat gland activity. A high GSR will typically indicate an increased cognitive load. The 5th reading will be measured during the cognitive task after physical fatigue.
Galvanic skin response (6th reading) | Periprocedural
  The electrical conductance of the skin, measured by Galvanic Skin Response (GSR), will be influenced by moisture levels resulting from sweat gland activity. A high GSR will typically indicate an increased cognitive load. The 6th reading will be measured after the cognitive task, after physical fatigue.
Nasa task load index | Periprocedural
  The different dimensions of task load, including mental demand, physical demand, temporal demand, performance, effort, and frustration, will be measured subjectively using the NASA Task Load Index (TLX). Low ratings will typically indicate an increased cognitive load. 1st reading will be taken after the cognitive task, before inducing physical fatigue.
Nasa task load index (2nd reading) | Periprocedural
  The different dimensions of task load, including mental demand, physical demand, temporal demand, performance, effort, and frustration, will be measured subjectively using the NASA Task Load Index (TLX). Low ratings will typically indicate an increased cognitive load. 2nd reading will be taken after the cognitive task, post physical fatigue induction.
Borg scale of perceived exertion | Periprocedural
  After achieving the mild intensity target heart rate range of 50-60% through treadmill training, the Borg Rate of Perceived Exertion (RPE) category scale (6-20) will be utilized to assess exertion levels. A higher score on this scale will indicate greater physical exertion.
Borg scale of perceived exertion (Ist reading) | Periprocedural
  Following the induction of physical fatigue, the Borg Rate of Perceived Exertion (RPE) category scale (6-20) will be used to evaluate exertion levels achieved during the treadmill training at the mild intensity target heart rate range of 50-60%. A higher score will reflect increased physical exertion. Ist reading will be taken after inducing physical fatigue.
Borg scale of perceived exertion (2nd reading) | Periprocedural
  After achieving the moderate intensity target heart rate range of 60-70% through treadmill training, the Borg Rate of Perceived Exertion (RPE) category scale (6-20) will be utilized to assess exertion levels. A higher score on this scale will indicate greater physical exertion. 2nd reading will be taken after the cognitive task prior to inducing physical fatigue.
Borg scale of perceived exertion (3rd reading) | Periprocedural
  Following the induction of physical fatigue, the Borg Rate of Perceived Exertion (RPE) category scale (6-20) will be used to evaluate exertion levels achieved during the treadmill training at the moderate intensity target heart rate range of 60-70%. A higher score will reflect increased physical exertion. 3rd reading will be taken after inducing physical fatigue.
Borg scale of perceived exertion (4rth reading) | Periprocedural
  After achieving the High-intensity target heart rate range of 70-80% through treadmill training, the Borg Rate of Perceived Exertion (RPE) category scale (6-20) will be utilized to assess exertion levels. A higher score on this scale will indicate greater physical exertion. 4rth reading will be taken after the cognitive task, before inducing physical fatigue.
Borg scale of perceived exertion (5th reading) | Periprocedural
  Following the induction of physical fatigue, the Borg Rate of Perceived Exertion (RPE) category scale (6-20) will be used to evaluate exertion levels achieved during the treadmill training at the High-intensity target heart rate range of 70-80%. A higher score will reflect increased physical exertion. 5th reading will be taken after inducing physical fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Imran Amjad, Phd, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No